CLINICAL TRIAL: NCT03479203
Title: Acute and Long-term Effects of E-Cigarette Aerosol Inhalation on Biomarkers of Endothelial Function and Vascular Reactivity
Brief Title: Acute Effects of E-Cigarette Aerosol Inhalation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Felix W. Wehrli, Professor of Radiologic Science, Biochemistry and Biophysics, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 828195; R01HL139358 (NIH)
Record Dates: First submitted 2018-02-28; First posted 2018-03-27 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Endothelial Dysfunction; Biochemical Markers
Keywords: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy, Non-Smokers (Experimental): Non-nicotinized electronic cigarette aerosol (16 2-second long puffs)
  Interventions: Drug: Electronic Cigarette Aerosol

INTERVENTIONS:
Drug: Electronic Cigarette Aerosol — 16 two-second-long puffs from a non-nicotinized electronic cigarette.

SUMMARY:
This study comprises a portion of a larger study designed to compare results of vascular function in non-smokers to vascular function in healthy smokers chronically exposed to nicotinized electronic cigarette aerosol versus conventional cigarettes.

DETAILED DESCRIPTION:
Here, we 1) investigate the acute effects of non-nicotinized e-cigarette aerosol inhalation in nonsmokers in terms of blood-based markers of inflammation and oxidative stress, and 2) evaluate their association with hemodynamic-metabolic MRI parameters quantifying peripheral vascular reactivity, cerebrovascular reactivity, and aortic stiffness.

ELIGIBILITY:
Inclusion Criteria:

• BMI of 18.5 - 30

Exclusion Criteria:

* Cancer
* HIV
* Mental illness
* Overt cardio- or neurovascular disease (prior heart attack, stroke, transient ischemic attacks)
* Serious arrhythmias
* Bronchospastic disease
* Upper respiratory tract infection within the past six weeks
* Chronic medication or antibiotics
* Claustrophobia / contraindications for MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix W. Wehrli, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zamani P, Proto EA, Wilson N, Fazelinia H, Ding H, Spruce LA, Davila A Jr, Hanff TC, Mazurek JA, Prenner SB, Desjardins B, Margulies KB, Kelly DP, Arany Z, Doulias PT, Elrod JW, Allen ME, McCormack SE, Schur GM, D'Aquilla K, Kumar D, Thakuri D, Prabhakaran K, Langham MC, Poole DC, Seeholzer SH, Reddy R, Ischiropoulos H, Chirinos JA. Multimodality assessment of heart failure with preserved ejection fraction skeletal muscle reveals differences in the machinery of energy fuel metabolism. ESC Heart Fail. 2021 Aug;8(4):2698-2712. doi: 10.1002/ehf2.13329. Epub 2021 May 15. PMID 33991175
- [Background] Langham MC, Caporale AS, Wehrli FW, Parry S, Schwartz N. Evaluation of Vascular Reactivity of Maternal Vascular Adaptations of Pregnancy With Quantitative MRI: Pilot Study. J Magn Reson Imaging. 2021 Feb;53(2):447-455. doi: 10.1002/jmri.27342. Epub 2020 Aug 25. PMID 32841482
- [Background] Kligerman S, Raptis C, Larsen B, Henry TS, Caporale A, Tazelaar H, Schiebler ML, Wehrli FW, Klein JS, Kanne J. Radiologic, Pathologic, Clinical, and Physiologic Findings of Electronic Cigarette or Vaping Product Use-associated Lung Injury (EVALI): Evolving Knowledge and Remaining Questions. Radiology. 2020 Mar;294(3):491-505. doi: 10.1148/radiol.2020192585. Epub 2020 Jan 28. PMID 31990264
- [Result] Chatterjee S, Caporale A, Tao JQ, Guo W, Johncola A, Strasser AA, Leone FT, Langham MC, Wehrli FW. Acute e-cig inhalation impacts vascular health: a study in smoking naive subjects. Am J Physiol Heart Circ Physiol. 2021 Jan 1;320(1):H144-H158. doi: 10.1152/ajpheart.00628.2020. Epub 2020 Nov 20. PMID 33216614
- [Result] Wehrli FW, Caporale A, Langham MC, Chatterjee S. New Insights From MRI and Cell Biology Into the Acute Vascular-Metabolic Implications of Electronic Cigarette Vaping. Front Physiol. 2020 May 21;11:492. doi: 10.3389/fphys.2020.00492. eCollection 2020. PMID 32528311
- [Result] Caporale A, Langham MC, Guo W, Johncola A, Chatterjee S, Wehrli FW. Acute Effects of Electronic Cigarette Aerosol Inhalation on Vascular Function Detected at Quantitative MRI. Radiology. 2019 Oct;293(1):97-106. doi: 10.1148/radiol.2019190562. Epub 2019 Aug 20. PMID 31429679
- [Result] Chatterjee S, Tao JQ, Johncola A, Guo W, Caporale A, Langham MC, Wehrli FW. Acute exposure to e-cigarettes causes inflammation and pulmonary endothelial oxidative stress in nonsmoking, healthy young subjects. Am J Physiol Lung Cell Mol Physiol. 2019 Aug 1;317(2):L155-L166. doi: 10.1152/ajplung.00110.2019. Epub 2019 May 1. PMID 31042077
- [Result] Caporale A, Lee H, Lei H, Rao H, Langham MC, Detre JA, Wu PH, Wehrli FW. Cerebral metabolic rate of oxygen during transition from wakefulness to sleep measured with high temporal resolution OxFlow MRI with concurrent EEG. J Cereb Blood Flow Metab. 2021 Apr;41(4):780-792. doi: 10.1177/0271678X20919287. Epub 2020 Jun 14. PMID 32538283

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy, Non-Smokers: Men and women between the ages of 18 and 35 years with no history of smoking, systemic disease, recent respiratory infection or chronic intake of medication.
Period: Overall Study
Arm/Group | Healthy, Non-Smokers
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pre-intervention status (i.e. pre-vaping).
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Information collected via self-reporting.
  Participants
    Hispanic or Latino | 2
    Not Hispanic or Latino | 29
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Blood-Based Biomarkers
Description: Post-vaping inflammation monitored by changes in an integrated cluster of blood-based biomarkers from serum/plasma of non-smoking healthy participants quantified at 0 and 120 min post-inhalation. The cluster consisted of: CRP, sICAM-1 in serum and HMGB1, ASC in plasma assayed using ELISA and quantified using absorbance-concentration curves generated by the manufacturers' standards; nitric oxide metabolites (nitrate + nitrite, NOx) in serum assayed with a nitrate/nitrite kit using a colorimetric standard provided by the manufacturer; reactive oxygen species (ROS) was quantified by using immortalized human pulmonary microvascular endothelial cells plated, prepared with serum, labeled with ROS dye and imaged confocal fluorescence microscopy.
  The outcome measure was expressed as fold increase over pre-vaping values.
Time Frame: Participant blood draws occurred at two time points: 1) pre-vaping, 2) 120 minutes post-vaping. Inflammation index is calculated from the fold change in biomarker values over pre-vaping values
Population: For each participant, the fold change is obtained as as logarithmic fold increases over pre-vaping values, as: log2(fold change) = log2(expression value(s) of post-vape biomarker) - log2(expression value(s) of pre-vape biomarker). Data are expressed as means ± SD (5 - 18 nanograms per milliliter range) and two-tailed paired t tests were used to determine statistical significance.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 31
fold change | 5 (0.5)
Statistical Analysis 1: Comparison: Healthy, Non-Smokers; Blood assessed for C-reactive protein (CRP), soluble intercellular adhesion molecule (sICAM), the high mobility group box-1 (HMGB1), the NLRP3 inflammasome, and nitrates (NOx for nitric oxide) pre- and post-vaping. CRP, sICAM HMGB1 and NLRP3 is in ng/ml blood and NOx is in nanomol/ml. These numbers were weighted to obtain an "inflammation index" in blood. This index represents the fold increase over pre-vaping values; Test type: Other — T-Test followed by Bonferroni post-hoc analysis; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [1 to 6], Standard Deviation 1.5

2. Primary Outcome: Acute Change in Aortic Pulse Wave Velocity Post-vaping
Description: Central arterial stiffness was assessed using aortic pulse-wave velocity (PWV), a biomarker of aortic stiffness calculated by measuring the velocity of a pulse wave between two points in the same artery. A higher aortic pulse wave velocity equates to a stiffer aorta.
  In each participant, aortic PWV was quantified, pre- and post-vaping, by dividing the path length of the aortic arch determined from a oblique sagittal image, by the transit time of the pulse pressure wave. Measurements obtained pre-vaping were compared to those obtained post-vaping.
Time Frame: PWV calculation occurred at two time points: 1) pre-vaping, 2) Fifteen minutes post-vaping.
Population: Participants* underwent an intervention which consisted of 16 3-second inhalations from a vaping device delivering non-nicotinized electronic cigarette aerosol. A quantitative magnetic resonance imaging scan was conducted pre- and post-vaping. Differences in aortic PWV before versus after e-cigarette vaping were assessed.
  *One participant not analyzed due to discomfort during the scan.
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 30
Meters per second | 0.19 (0.20)

3. Primary Outcome: Change in Femoral Artery Flow-Mediated Dilation Post-Vaping
Description: Degree of dilation (% change in cross-sectional area) of femoral artery during hyperemia (the transient increase in blood flow velocity) after e-cigarette vaping as compared to before e-cigarette vaping.
Time Frame: Flow mediated dilation calculation occurred at two time points: 1) pre-vaping, 2) 40 minutes post-vaping.
Population: Participants* underwent an intervention which consisted of 16 3-second inhalations from a vaping device delivering non-nicotinized electronic cigarette aerosol. A quantitative magnetic resonance imaging scan was conducted pre- and post-vaping. Differences in flow mediated dilation before versus after e-cigarette vaping were assessed.
  *One participant not analyzed due to discomfort during the scan.
Measure: Mean (Standard Deviation); unit: percentage of change in cross-sectional
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 30
percentage of change in cross-sectional | -3.20 (0.90)

4. Primary Outcome: Change in Washout Time Post-Vaping
Description: Transit time of desaturated capillary blood from tissue to the imaging location after e-cigarette vaping
Time Frame: Washout time calculation occurred at two time points: 1) pre-vaping, and 2) 40 minutes post-vaping
Population: Participants underwent an intervention which consisted of 16 3-second inhalations from a vaping device delivering non-nicotinized electronic cigarette aerosol. A 50 minute quantitative magnetic resonance imaging protocol was conducted pre- and immediately post-vaping. (One participant not analyzed due discomfort with the cuff occlusion portion of the protocol.)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 30
Seconds | -1.50 (0.30)

5. Primary Outcome: Change in Upslope Post-Vaping
Description: Tissue oxygen resaturation rate after e-cigarette vaping.
Time Frame: Upslope was calculated at two time points: 1) pre-vaping, and 2) 40 minutes post-vaping
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation/sec
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 30
percentage of oxygen saturation/sec | 0 (0.20)

6. Primary Outcome: Change in Overshoot Post-Vaping
Description: Degree of overcompensatory effect post-vaping in the supply of oxygen after ischemia.
Time Frame: Overshoot was calculated at two time points: 1) pre-vaping, and 2) 40 minutes post-vaping.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation/sec
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 30
percentage of oxygen saturation/sec | 10 (2.0)

7. Primary Outcome: Change in Breath Hold Index Post-Vaping
Description: Rate of increase in blood flow velocity in the superior sagittal sinus from intermittent volitional apnea.
Time Frame: Breath hold index was calculated at two time points: 1) pre-vaping, 2) five minutes post-vaping.
Population: Participants underwent an intervention which consisted of 16 3-second inhalations from a vaping device delivering non-nicotinized electronic cigarette aerosol. A 50 minute quantitative magnetic resonance imaging protocol was conducted pre- and post-vaping. (One participant not analyzed due discomfort with the cuff occlusion portion of the protocol.)
Measure: Mean (Standard Deviation); unit: Centimeters per Seconds Squared
Arm/Group | Healthy, Non-Smokers
Number analyzed (Participants) | 30
Centimeters per Seconds Squared | -0.02 (0.02)

ADVERSE EVENTS:
Time Frame: Six Hours.
Arm/Group | Healthy, Non-Smokers
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03479203/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT03479203/ICF_001.pdf